CLINICAL TRIAL: NCT06131450
Title: A Phase Ib/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of BL-M07D1 for Injection in Patients With HER2-expressing Recurrent or Metastatic Gynecologic Malignancies
Brief Title: A Study of BL-M07D1 in Patients With HER2-expressing Recurrent or Metastatic Gynecologic Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-203
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Gynecological Malignancies
Keywords: HER2 expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-M07D1 (Experimental): Participants receive BL-M07D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M07D1

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion

SUMMARY:
This study is a single-arm, open, multicenter, non-randomized phase Ib/II clinical study evaluating the efficacy and safety of BL-M07D1 for injection in patients with HER2-expressing recurrent or metastatic gynecologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Female;
3. Age: ≥18 years old and ≤75 years old;
4. Expected survival time ≥3 months;
5. patients with recurrent or metastatic HER2-positive/low-expression gynecologic malignancies who have failed or are intolerant to standard treatment or who currently have no standard treatment;
6. The histopathology of gynecological malignant tumors should meet the following conditions: HER2 positive; Low expression of HER2;
7. Consent to provide archived tumor tissue samples or fresh tissue samples of primary or metastatic lesions within 2 years;
8. At least one measurable lesion meeting the RECIST v1.1 definition was required;
9. ECOG score 0 or 1;
10. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 defined by NCI-CTCAE v5.0;
11. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
12. No blood transfusion, use of any cell growth factors and/or platelet-raising drugs were allowed within 14 days before screening, and the organ function level had to be acceptable;
13. Urinary protein ≤2+ or ≤1000mg/24h;
14. albumin ≥30 g/L;
15. Women who are likely to give birth must have negative serum/urine pregnancy within 7 days before treatment and must be non-lactating; All enrolled patients should have adequate contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. had received anti-tumor therapy before the first dose; Mitomycin and nitrosoureas; Oral fluorouracils; Palliative radiotherapy; Anti-tumor traditional Chinese medicine or Chinese patent medicine;
2. had received prior ADC drug therapy with camptothecin derivative (topoisomerase I inhibitor) as toxin;
3. had a history of serious cardiovascular and cerebrovascular diseases;
4. active autoimmune or inflammatory diseases;
5. Patients with other malignant tumors within 5 years before the first administration, except cured skin squamous cell carcinoma, basal cell carcinoma, superficial bladder cancer and prostate/cervix/breast cancer in situ;
6. Unstable thrombotic events such as deep vein thrombosis, arterial thrombosis, and pulmonary embolism requiring medical intervention within 6 months before screening;
7. patients with massive or symptomatic effusions or poorly controlled effusions;
8. Hypertension poorly controlled by antihypertensive drugs (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
9. Current interstitial lung disease, drug-induced interstitial pneumonia, radiation pneumonitis requiring steroid therapy, or a history of these diseases;
10. patients with central nervous system (CNS) metastases and/or carcinomatous meningitis (meningeal metastases);
11. patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any ingredient of BL-M07D1;
12. patients received previous organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
13. HIVAb positive, active tuberculosis, active hepatitis B virus infection, or active hepatitis C virus infection;
14. active infections requiring systemic therapy, such as severe pneumonia, bacteremia, sepsis, etc.;
15. had participated in another clinical trial within 4 weeks before the first dose;
16. pregnant or lactating women;
17. The investigator did not consider it appropriate to apply other criteria for participation in the trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M07D1.
Phase II: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M07D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1.
Phase Ib: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Progression-free Survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of BL-M07D1 to the first date of either disease progression or death, whichever occurs first.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-M07D1 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-M07D1 will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-M07D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-BL-M07D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, PHD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China